CLINICAL TRIAL: NCT00061464
Title: ALIMTA Plus Gemcitabine as Front-Line Chemotherapy for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Phase II Clinical Trial
Brief Title: Pemetrexed Plus Gemcitabine for Patients With Locally Advanced or Metastatic NSCLC Who Have Not Had Previous Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7211; H3E-US-JMFX
Record Dates: First submitted 2003-05-28; First posted 2003-05-29 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: pemetrexed
Drug: gemcitabine

SUMMARY:
The purposes of this study are to determine:

1. The safety of pemetrexed plus Gemcitabine and any side effects that might be associated with the combination of these two drugs.
2. Whether pemetrexed plus Gemcitabine can help patients with non-small cell lung cancer live longer.
3. Whether pemetrexed plus Gemcitabine can make the tumor smaller or disappear, and for how long.
4. To see if patients feel better while taking pemetrexed plus Gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Non-Small Cell Lung Cancer that can be treated with chemotherapy
* Have received no prior chemotherapy for Non-Small Cell Lung Cancer
* Have at least one measurable lesion
* Have an adequate performance status
* Sign an informed consent

Exclusion Criteria:

* A female who is pregnant or breastfeeding
* Treatment with an investigational drug within the last 30 days, previously completed or withdrawn from this study or any other study investigating pemetrexed
* Treatment with radiation therapy within the last 1-2 weeks
* Brain metastasis that is uncontrolled
* Active infection or other serious condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-02; Study Completion 2006-02

PRIMARY OUTCOMES:
To determine the tumor response rate for pemetrexed plus gemcitabine in patients with locally advanced or metastatic (Stage IIIB or IV) Non-Small Cell Lung Cancer (NSCLC).

SECONDARY OUTCOMES:
To measure time-to-event efficacy variables including:
time to objective tumor response for responding patients
duration of response for responding patients
time to treatment failure
time to progressive disease
progression-free survival
overall survival
To characterize the quantitative and qualitative toxicities of pemetrexed plus gemcitabine in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Columbia, South Carolina